CLINICAL TRIAL: NCT06494267
Title: The Effect of Video-Assisted Self-Assessment on Nasogastric Tube Insertion Knowledge and Skills: A Randomized Controlled Trial
Brief Title: Video-Assisted Self-Assessment on Nasogastric Tube Insertion
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Bahar Ciftci, Principal Investigator, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Toplantı/Karar Sayısı:8 /3
Record Dates: First submitted 2024-07-02; First posted 2024-07-10 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Nurse's Role

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Students will be videotaped while performing a nasogastric tube placement and will be asked to make a self-assessment.
  Interventions: Behavioral: Experimental (Video-Assisted Self-Assessment on Nasogastric Tube Insertion)
- Control (No Intervention): No application will be made.

INTERVENTIONS:
Behavioral: Experimental (Video-Assisted Self-Assessment on Nasogastric Tube Insertion) — Students in the experimental group will be videotaped while practicing and students will make self-evaluations.
  Arms: Experimental

SUMMARY:
Introduction and Purpose Advancements in Nursing Education: The integration of technology, specifically video-supported training, is a significant development in nursing education.

Focus on Nasogastric Tube (NGT) Placement: Proper placement of NGT is a critical skill in nursing. Traditional methods alone may not suffice in acquiring and maintaining this skill.

Objective: Evaluate the impact of video-supported self-assessment on the knowledge and skills of nursing students regarding NGT placement.

Hypotheses Video-supported self-assessment increases students' knowledge about NGT placement.

Video-supported self-assessment enhances students' skills in NGT placement. Materials and Methods Design: A randomized controlled pre-test and post-test experimental design. Ethics: Ethical approval will be obtained and registered with Clinical Trials ID.

Data Collection Tools:

FR.1 Personal Information Form: Demographic data collection. FR.2 NGT Placement Knowledge Test: 20 multiple-choice questions based on theoretical content.

FR.3 NGT Placement Skill Checklist: 51 steps evaluating correct, incorrect, and unobserved applications.

Data Collection Process Initial Phase: Explanation of the study, informed consent, and completion of the FR.1 form and FR.2 pre-test.

Traditional Teaching: A theoretical lecture on NGT placement.

Practical Application:

Experimental Group: Practical demonstration recorded and shared with students for self-assessment.

Control Group: Practical demonstration recorded but not shared with students. Post-Intervention Assessment: FR.2 post-test and an OSCE exam based on FR.3 for both groups after one week.

Data Analysis Software: SPSS 23.0. Methods: T-tests, Chi-square tests, Pearson and Spearman correlation analyses depending on data distribution.

Statistical Significance: p<0.05. Study Limitations Scope: Limited to first-year nursing students at one university. Interaction: Potential interaction between intervention and control group students.

Ethical Principles Approval: Obtained from the Ethics Committee and the university. Participant Rights: Informed consent, respect for autonomy, confidentiality, and adherence to the Helsinki Declaration.

This summary captures the essence of the research study described in the original document, focusing on the purpose, methods, data collection, analysis, limitations, and ethical considerations.

DETAILED DESCRIPTION:
Introduction and Purpose Today, with the advancement of technology, the diversification of methods used in nursing education is an important development. Video-assisted education stands out among these developments. Video-assisted education is considered an effective tool for improving nurses' clinical skills and ensuring their correct application. Nasogastric tube (NGT) insertion skill is a basic ability in nursing practice and its correct performance is of vital importance. However, acquisition and maintenance of this skill may not be sufficient by traditional education methods alone. In this context, video-assisted self-assessment may play an important role in the assessment of NGS insertion knowledge and skill in nursing education. The aim of this study is to evaluate the effect of video-assisted self-assessment on nasogastric tube insertion knowledge and skill in nursing clinical skills education. Hypotheses The use of video-assisted self-assessment method increases students' knowledge level regarding nasogastric tube insertion practice. The use of video-assisted self-assessment method increases students' skill level regarding nasogastric tube insertion practice. Material and Method This research was designed as a randomized controlled pretest-posttest experimental design. Since the study is a randomized controlled trial, the Clinical Trials ID will be obtained after the ethics committee is approved. The Intervention Description and Replication Template (TIDier) checklist and guide were used to define the intervention. "FR.1 Personal Information Form", "FR.2 Nasogastric Tube Placement Knowledge Test" and "FR.3 Nasogastric Tube Placement Skills Checklist" will be used to collect data. Data Collection Tools FR.1 Personal Information Form: It was prepared by the researchers and consists of 15 questions questioning demographic characteristics such as age, gender, and socioeconomic level. FR.2 Nasogastric Tube Placement Knowledge Test: A knowledge test was created in line with the scope and objectives of the NGS placement theoretical course content prepared in line with the literature. It consists of 20 multiple-choice questions with five options. The lowest score possible from this test is 0 and the highest is 20. FR.3 Nasogastric Tube Placement Skill Checklist: It includes the materials to be used in the NGS placement application and the steps to ensure that the application is carried out correctly. It consists of 51 steps. Each procedure step will be evaluated and scored as "Correct Application", "Incorrect Application" and "Not Observed". Data Collection Data will be collected in the Fundamentals of Nursing course in the spring semester of the 2023-2024 academic year. In the first stage, all students will be informed about the research and their consent will be obtained. Students who agree to participate in the research will fill out the "FR.1 Personal Information Form" in the classroom. Then, all students will be given the "FR.2 Knowledge Test for Nasogastric Tube Placement" as a pretest. Experimental and Control Groups Experimental Group: Students will be shown the NGS placement application in a laboratory environment and will be applied on a model. All procedures will be recorded with a fixed camera and their own video recordings will be sent to the students. Students will be asked to watch the videos and evaluate them according to the application skill list. Control Group: Students will be shown the NGS placement application in a laboratory environment and will be applied on a model. All procedures will be recorded with a fixed camera, but the recordings will not be shared with the students. Post-Test and OSCE The "FR.2 Nasogastric Tube Placement Knowledge Test" will be applied as a post-test to the students in the experimental and control groups one week after the completion of theoretical training and laboratory practice. At the same time, the OSCE exam will be performed in accordance with the FR.3 checklist for both groups. Data Evaluation SPSS 23.0 package program will be used to evaluate the data obtained from the research. The suitability of the variables for normal distribution will be examined with visual and analytical methods. Independent groups t-test and chi-square test will be used for comparisons of the control and intervention groups. Paired t test or Wilcoxon test will be used to compare the scale scores before and after the application in the intervention group. The relationships between the variables will be evaluated with Pearson or Spearman correlation analysis. The level of statistical significance will be accepted as p<0.05. Difficulties and Limitations of the Study This study was conducted only with first-year nursing students studying at the faculty of nursing of a university. Additionally, the possibility of interaction between the students in the intervention and control groups increases the limitations of the study. Ethical Principles of the Study Before starting the research, approval will be obtained from the Ethics Committee Presidency. In addition, written permission will be obtained from the university where the research will be conducted. During the collection of research data, individuals will be informed about the research and the "Informed Consent" principle will be fulfilled, stating that they are free to participate or not in the research, the "Respect for Autonomy" principle, and stating that the participants' information will be kept confidential, and written and verbal consent will be obtained. Since individual rights must be protected in the research, the Helsinki Declaration of Human Rights will be adhered to.

ELIGIBILITY:
Inclusion Criteria:

* Being 18 years of age or older
* Being a first-year student at the Faculty of Nursing
* Being taking the Fundamentals of Nursing course for the first time
* Not coming as a horizontal or vertical transfer
* Not being absent on the dates when the research data will be collected
* Being willing to participate in the research and giving written consent

Exclusion Criteria:

* Those who are not first-year nursing students
* Students who come via horizontal or vertical transfer
* Students who graduated from Health Vocational High School
* Students in the intervention group who are not subject to video-assisted self-assessment method
* Students who want to leave the study for any reason during the research process

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 65 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-09-10 (Estimated)

PRIMARY OUTCOMES:
FR.1 Personal Information Form: | 3months
  This form was prepared by the researchers and consists of 15 questions questioning the demographic characteristics of the students such as age, gender, socioeconomic level, etc.

SECONDARY OUTCOMES:
FR.2 Nasogastric Tube Placement Knowledge Test: | 3months
  A knowledge test was created by the researcher in line with the scope and objectives of the theoretical course content of NGS placement prepared in line with the literature (Lynn, P. (2018)). The knowledge test consists of 20 multiple-choice questions with five options that question the information required for NGS placement. The lowest score possible from this test is 0 (zero), and the highest is 20. The distribution of questions in the knowledge test was prepared according to the target behaviors within the subject.

OTHER OUTCOMES:
FR.3 Nasogastric Tube Placement Skill Checklist: | 3months
  It includes the materials to be used in the Nasogastric Tube Placement application and the steps to ensure that the application is carried out correctly. The checklist prepared by the researcher consists of 51 steps. Each procedure step will be evaluated as "Correct Application", "Incorrect Application" and "Not Observed" and each will be scored considering the characteristics of the procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Bahar Çiftçi, Study Director — Ataturk University
Locations (1):
- Atatürk University Faculty of Nursing, Erzurum, Turkey (Türkiye)

REFERENCES:
- [Derived] Yavuz B, Koc G, Yuce Basaran HD, Ciftci B. Watch and learn your performance: The effect of self-assessment with video recording on nursing students' knowledge and skills of nasogastric catheter placement-A randomized controlled trial. Nurse Educ Pract. 2025 Feb;83:104251. doi: 10.1016/j.nepr.2025.104251. Epub 2025 Jan 10. PMID 39826351